CLINICAL TRIAL: NCT05559437
Title: Ultrasound-guided Ilioinguinal/Iliohypogastric Nerve Block Compared to Posterior Quadratus Lumborum Block in Patients Undergoing Inguinal Hernia Repair
Brief Title: Ultrasound-guided Ilioinguinal/Iliohypogastric Nerve Block
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mona Gad
Record Dates: First submitted 2022-09-24; First posted 2022-09-29 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Inguinal Hernia Repair; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: To investigate the effectiveness of ultrasound guided Ilioinguinal/Iliohypogastric ( II/IH) block compared to ultrasound guided Posterior Quadratus Lumborum (PQL) block in patients subjected to inguinal hernia repair.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum Block group (Experimental): Quadratus lumborum group (Q) (n=30): patients will receive Quadratus Lumborum Block using 20 mL of 0.25% Levo-bupivacaine
  Interventions: Drug: Levo-bupivacaine 0.25
- Ilioinguinal/Iliohypogastric Nerve Block group (Experimental): Ilioinguinal/Iliohypogastric Nerve Block group (I) (n=30): patients will receive Ilioinguinal/Iliohypogastric Nerve Block using 5 mL of 0.25%Levo- bupivacaine
  Interventions: Drug: Levo-bupivacaine 0.25

INTERVENTIONS:
Drug: Levo-bupivacaine 0.25 — The blockade of ilioinguinal/iliohypogastric nerves in the anterior abdominal wall has improved postoperative analgesia after open inguinal hernia repair. Other new blocks needs to be investigated

SUMMARY:
Abdominal wall hernias are common, with a prevalence of 1.7% for all ages and 4% for those aged over 45 years. Inguinal hernias account for 75% of abdominal wall hernias, with a lifetime risk of 27% in men and 3% in women. Repair of inguinal hernia is one of the most common operations in general surgery

DETAILED DESCRIPTION:
The peripheral nerve block usage is increasing in popularity because it decreases pain as estimated by visual analogue scores/numerical rating pain scores postoperatively and decreases the need for postoperative analgesic usage thereby reducing opioid induced side effects like postoperative respiratory depression, nausea, vomiting, NSAID induced gastritis etc. Nerve blocks also shorten Post-Anesthesia Care Unit stay time, and also increases patient satisfaction .

Ultrasound-guided peripheral nerve blocks including ilioinguinal/ iliohypogastric nerve block and transversus abdominis plane block have been widely used and considered as effective traditional techniques for postoperative analgesia in inguinal hernia repair .

In recent years, the quadratus lumborum (QL) block is proposed to be an alternative regional block for both upper abdominal surgery and lower abdominal surgery.

The blockade of ilioinguinal/iliohypogastric nerves in the anterior abdominal wall has improved postoperative analgesia after open inguinal hernia repair and many other procedures.

The Quadratus Lumborum (QL) Block is a regional anesthetic technique which described by anesthesiologist "DR Rafael Blanco" in 2007. Quadratus Lumborum block allows the local anesthetic agent to spread between the posterior aspect of the Quadratus Lumborum muscle and the middle layer of the Thoracolumbar fascia, which is nearer to the thoracic paravertebral space. It has four approaches based on the point of drug deposition in relation to quadratus lumborum muscle. Drug is deposited on the anterolateral, posterior, anterior to the Quadratus Lumborum muscle in the three approaches. In fourth approach drug is deposited intramuscularly. It provides postoperative analgesia for longer duration .

ELIGIBILITY:
Inclusion Criteria:

1. all patients undergoing elective or emergent unilateral inguinal hernia repair
2. Patients scheduled for unilateral inguinal hernia repair

Exclusion Criteria:

1. Patient refusal.
2. Contraindication to neuraxial block.
3. neuromuscular diseases (as myopathies, myasthenia gravies).
4. Hematological diseases, bleeding or coagulation abnormality.
5. Uncontrolled Psychiatric diseases,
6. Local skin infection and sepsis at site of the block.
7. Known intolerance to the study drugs.
8. Body Mass Index > 40 Kg/m2,
9. Unstable cardiovascular condition

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Post Operative Pain | 0 hour after the operation up to 24-hour analgesic after surgery
  All patients will be familiar with the use of the visual analogue scale score identifying 0 as no pain and 10 as worst imaginable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Gad, Assist.Prof, Principal Investigator — Department of anesthesia and SICU,Faculty of medicine,Mansoura university , Egypt.
Locations (1):
- Mansoura university Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided